CLINICAL TRIAL: NCT02580552
Title: A Phase 1 Dose-ranging Study to Investigate the Safety, Tolerability, and Pharmacokinetics of MRG-106 Following Local Intratumoral, Subcutaneous, and Intravenous Administration in Subjects With Various Lymphomas and Leukemias
Brief Title: Safety, Tolerability and Pharmacokinetics of MRG-106 in Patients With Mycosis Fungoides (MF), CLL, DLBCL or ATLL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: miRagen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRG106-11-101
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Cutaneous T-cell Lymphoma (CTCL); Mycosis Fungoides (MF); Chronic Lymphocytic Leukemia (CLL); Diffuse Large B-Cell Lymphoma (DLBCL), ABC Subtype; Adult T-Cell Leukemia/Lymphoma (ATLL)
Keywords: Cutaneous T-cell Lymphoma; CTCL; Mycosis Fungoides; Chronic lymphocytic leukemia; CLL; Diffuse large B-cell lymphoma; DLBCL; Adult T-cell leukemia/lymphoma; ATLL
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia-Lymphoma, Adult T-Cell | interventions — cobomarsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A, MF (Experimental): Intratumoral Injection of cobomarsen
  Interventions: Drug: Cobomarsen
- Part B, MF (Experimental): Subcutaneous, intravenous or a combination of systemic and intratumoral administration of cobomarsen with or without stable background therapy
  Interventions: Drug: Cobomarsen
- Part C, MF (Experimental): Subcutaneous or intravenous administration of cobomarsen as monotherapy
  Interventions: Drug: Cobomarsen
- Part D, CLL (Experimental): Subcutaneous or intravenous administration of cobomarsen as monotherapy
  Interventions: Drug: Cobomarsen
- Part E, DLBCL, activated B-cell (ABC) subtype (Experimental): Subcutaneous or intravenous administration of cobomarsen as monotherapy
  Interventions: Drug: Cobomarsen
- Part F, ATLL (Experimental): Subcutaneous or intravenous administration of cobomarsen as monotherapy
  Interventions: Drug: Cobomarsen

INTERVENTIONS:
Drug: Cobomarsen
  Other Names: MRG-106

SUMMARY:
Objectives of this clinical trial are to evaluate the safety, tolerability, pharmacokinetics and potential efficacy of the investigational drug, cobomarsen (MRG-106), in patients diagnosed with certain lymphomas and leukemias, including cutaneous T-cell lymphoma (CTCL) [mycosis fungoides (MF) subtype], chronic lymphocytic leukemia (CLL), diffuse large B-cell lymphoma (DLBCL) [activated B-cell (ABC) subtype], and adult T-cell leukemia/lymphoma (ATLL). Cobomarsen is an inhibitor of a molecule called miR-155 that is found at high levels in these types of cancers and may be important in promoting the growth and survival of the cancer cells. Participants in the clinical trial will receive weekly doses of cobomarsen administered by injection under the skin or into a vein, or by injection directly into cancerous lesions in the skin (for CTCL only). Blood samples will be collected to measure how cobomarsen is processed by the body, and other measurements will be performed to study how normal and cancerous cells of the immune system respond when exposed to cobomarsen.

DETAILED DESCRIPTION:
Study Design:

* Part A: Cohorts of 3-6 patients diagnosed with MF will receive up to five intratumoral injections of cobomarsen over a period of up to 15 days with follow-up for an additional 20 days, beginning with the maximum deliverable intratumoral dose. Doses may be decreased in subsequent cohorts to determine the minimum pharmacodynamically active dose.
* Parts B-F: Patients in these parts of the study will be diagnosed with MF (Parts B and C), CLL (Part D), DLBCL (Part E), or ATLL (Part F). All patients will receive subcutaneous or intravenous cobomarsen (or a combination of systemic and intratumoral administration for MF patients only) on Days 1, 3 and 5, and will continue dosing on a weekly schedule until the patient becomes intolerant, develops clinically significant side effects, progresses, or the trial is terminated. Doses administered will not exceed a dose level predicted to be safe based on all prior treatment experience with the drug. Patients in Part B may continue on a stable background therapy for their disease during their treatment with cobomarsen, while patients in Parts C-F will be treated with cobomarsen alone.

ELIGIBILITY:
Inclusion Criteria:

* Parts A-C only: Patients must have biopsy proven MF, clinical stage I, II, or III (excluding visceral or nodal involvement), and must be refractory to or intolerant of established therapies for their condition
* Part D only: Patients diagnosed with CLL who are intolerant to, or have disease that is relapsed/refractory after, at least two prior therapies
* Part E only: Patients with biopsy-proven DLBCL who are intolerant to, or have disease that is relapsed/refractory after, at least two prior therapies, including any anti-CD20 monoclonal antibody and chemotherapy with curative intent
* Part F only: Patients with documented HTLV-1 infection and histologically or cytologically proven ATLL of any stage, and who are intolerant to, or have disease that is relapsed/refractory after, at least one prior therapy
* Females must not be pregnant or lactating. Women of child-bearing potential must use a highly effective method of contraception throughout their study participation and for at least 6 months following the last dose of study drug.
* Males must be surgically sterile, abstinent, or if engaged in sexual relations with a female of child-bearing potential, must be willing to use a highly effective method of contraception throughout their study participation and for at least 6 months after the last dose of study drug.

Exclusion Criteria:

* Evidence of renal or liver dysfunction at screening
* Clinically significant anemia, neutropenia or thrombocytopenia at screening
* History of bleeding diathesis or coagulopathy
* Clinically significant cardiovascular disease, history of myocardial infarction within the last 6 months, or evidence of QTc interval prolongation at screening
* Serologically positive for HIV; serologically positive for Hepatitis B or Hepatitis C with evidence of liver dysfunction or documented liver cirrhosis
* Prior malignancies within the past 3 years (with allowance for adequately treated in situ carcinoma of the cervix uteri, and basal cell or localized squamous cell carcinoma of the skin treated with curative intent)
* Use of an investigational small molecule drug during the 30 days prior to screening or use of an investigational oligonucleotide or biologic drug during the prior 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of cobomarsen based on vital signs, physical examination, clinical laboratory tests, ECG, and incidence and severity of adverse events | From start of treatment to end of study participation

SECONDARY OUTCOMES:
Area under the plasma concentration vs. time curve (AUC) of cobomarsen following single and repeat doses administered intratumorally, subcutaneously or intravenously | Up to 56 days
Peak plasma concentration (Cmax) of cobomarsen following single and repeat doses administered intratumorally, subcutaneously or intravenously | Up to 56 days
Trough plasma concentration (Ctrough) of cobomarsen following each 4-week cycle of dosing | Monthly from Week 5 up to end of study participation
Skin disease severity (index lesions) - MF only | Every 2 weeks from start of treatment until end of study participation
  Changes in MF skin lesion severity before and after treatment based on the Composite Assessment of Index Lesion Severity (CAILS) score
Skin disease severity (whole body) - MF only | Every 2 weeks from start of treatment until end of study participation
  Changes in MF skin lesion severity before and after treatment based on the modified Severity Weighted Assessment Tool (mSWAT) score
Overall Response Rate in the skin - MF | Approximately 1 year
  Proportion of subjects who achieve a partial response (PR) or complete response (CR) in the skin, based on SWAT score
Overall Response Rate - CLL | Approximately 1 year
  Proportion of subjects who achieve a PR or CR as defined by IWCLL criteria (Hallek et al., 2008) based on CT scans, bone marrow biopsies, and flow cytometry
Minimal Residual Disease (MRD) - CLL only | Approximately 1 year
  Proportion of subjects who achieve a CR with no evidence of MRD by flow cytometry
Overall Response Rate - DLBCL | Approximately 1 year
  Proportion of subjects who achieve a PR or CR as defined by the Lugano classification (Cheson et al., 2014) based on positron emission tomography-computed tomography (PET-CT) scans and bone marrow biopsy to confirm CR
Overall Response Rate - ATLL | Approximately 1 year
  Proportion of subjects who achieve a PR or CR as defined by international consensus criteria (Tsukasaki et al., 2009) based on CT scans and flow cytometry, and bone marrow biopsy to confirm CR
Duration of Response | Up to approximately 2 years
  Number of days from initial date of confirmed PR or CR until loss of response or relapse
Time to Progression | Up to approximately 2 years
  Number of days from first dose until objective disease progression
Progression Free Survival (PFS) | Up to approximately 2 years
  Number of days from first dose until objective disease progression or death from any cause
Overall Survival (OS) | Up to approximately 2 years
  Number of days from first dose until death from any cause

OTHER OUTCOMES:
miR-155-5p expression in cutaneous lesions of subjects with MF | At baseline and between Week 16 and end of study participation
  Exploratory assessment based on quantitative real time polymerase chain reaction (qRT-PCR) analysis of total RNA isolated from skin biopsies
Proportion of neoplastic lymphoid cells in cutaneous lesions of subjects with MF | At baseline and between Week 16 and end of study participation
  Exploratory histological assessment before and after treatment with cobomarsen
Proportions of immune cell subsets | At baseline and monthly or bimonthly, up to end of study participation
  Exploratory assessment before and after treatment with cobomarsen by flow cytometry on whole blood
Dermatology-specific quality of life - MF only | At baseline and monthly, up to approximately 2 years
  Changes in skin-related quality of life based on the Skindex-29 assessment tool
Pruritus - MF only | At baseline and monthly, up to approximately 2 years
  Changes in intensity of skin itch based on the Pruritus Numerical Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Diana M. Escolar, MD, FAAN, Study Director — miRagen Therapeutics, Inc.
Locations (19):
- United States (19):
  - City of Hope, Duarte, California
  - UCSD Moores Cancer Center, La Jolla, California
  - UCLA Department of Medicine, Los Angeles, California
  - Chao Family Comprehensive Cancer Center at University of California, Irvine, Orange, California
  - Stanford University Hospital and Clinics, Stanford, California
  - University of Colorado, Anschutz Medical Campus, Aurora, Colorado
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northwestern University; Department of Dermatology, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Inova Melanoma and Skin Cancer Center / Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Kester MS, Ballabio E, Benner MF, Chen XH, Saunders NJ, van der Fits L, van Doorn R, Vermeer MH, Willemze R, Tensen CP, Lawrie CH. miRNA expression profiling of mycosis fungoides. Mol Oncol. 2011 Jun;5(3):273-80. doi: 10.1016/j.molonc.2011.02.003. Epub 2011 Feb 24. PMID 21406335
- [Background] Moyal L, Barzilai A, Gorovitz B, Hirshberg A, Amariglio N, Jacob-Hirsch J, Maron L, Feinmesser M, Hodak E. miR-155 is involved in tumor progression of mycosis fungoides. Exp Dermatol. 2013 Jun;22(6):431-3. doi: 10.1111/exd.12161. PMID 23711069
- [Background] Maj J, Jankowska-Konsur A, Sadakierska-Chudy A, Noga L, Reich A. Altered microRNA expression in mycosis fungoides. Br J Dermatol. 2012 Feb;166(2):331-6. doi: 10.1111/j.1365-2133.2011.10669.x. Epub 2012 Jan 9. PMID 21966986
- [Background] Kopp KL, Ralfkiaer U, Gjerdrum LM, Helvad R, Pedersen IH, Litman T, Jonson L, Hagedorn PH, Krejsgaard T, Gniadecki R, Bonefeld CM, Skov L, Geisler C, Wasik MA, Ralfkiaer E, Odum N, Woetmann A. STAT5-mediated expression of oncogenic miR-155 in cutaneous T-cell lymphoma. Cell Cycle. 2013 Jun 15;12(12):1939-47. doi: 10.4161/cc.24987. Epub 2013 May 15. PMID 23676217
- [Background] Eis PS, Tam W, Sun L, Chadburn A, Li Z, Gomez MF, Lund E, Dahlberg JE. Accumulation of miR-155 and BIC RNA in human B cell lymphomas. Proc Natl Acad Sci U S A. 2005 Mar 8;102(10):3627-32. doi: 10.1073/pnas.0500613102. Epub 2005 Feb 28. PMID 15738415
- [Background] Cui B, Chen L, Zhang S, Mraz M, Fecteau JF, Yu J, Ghia EM, Zhang L, Bao L, Rassenti LZ, Messer K, Calin GA, Croce CM, Kipps TJ. MicroRNA-155 influences B-cell receptor signaling and associates with aggressive disease in chronic lymphocytic leukemia. Blood. 2014 Jul 24;124(4):546-54. doi: 10.1182/blood-2014-03-559690. Epub 2014 Jun 9. PMID 24914134
- [Background] Guinn D, Ruppert AS, Maddocks K, Jaglowski S, Gordon A, Lin TS, Larson R, Marcucci G, Hertlein E, Woyach J, Johnson AJ, Byrd JC. miR-155 expression is associated with chemoimmunotherapy outcome and is modulated by Bruton's tyrosine kinase inhibition with Ibrutinib. Leukemia. 2015 May;29(5):1210-3. doi: 10.1038/leu.2014.344. Epub 2014 Dec 9. No abstract available. PMID 25486872
- [Background] Tomita M. Important Roles of Cellular MicroRNA miR-155 in Leukemogenesis by Human T-Cell Leukemia Virus Type 1 Infection. ISRN Microbiol. 2012 Sep 18;2012:978607. doi: 10.5402/2012/978607. Print 2012. PMID 23762762
- [Background] Olsen EA, Whittaker S, Kim YH, Duvic M, Prince HM, Lessin SR, Wood GS, Willemze R, Demierre MF, Pimpinelli N, Bernengo MG, Ortiz-Romero PL, Bagot M, Estrach T, Guitart J, Knobler R, Sanches JA, Iwatsuki K, Sugaya M, Dummer R, Pittelkow M, Hoppe R, Parker S, Geskin L, Pinter-Brown L, Girardi M, Burg G, Ranki A, Vermeer M, Horwitz S, Heald P, Rosen S, Cerroni L, Dreno B, Vonderheid EC; International Society for Cutaneous Lymphomas; United States Cutaneous Lymphoma Consortium; Cutaneous Lymphoma Task Force of the European Organisation for Research and Treatment of Cancer. Clinical end points and response criteria in mycosis fungoides and Sezary syndrome: a consensus statement of the International Society for Cutaneous Lymphomas, the United States Cutaneous Lymphoma Consortium, and the Cutaneous Lymphoma Task Force of the European Organisation for Research and Treatment of Cancer. J Clin Oncol. 2011 Jun 20;29(18):2598-607. doi: 10.1200/JCO.2010.32.0630. Epub 2011 May 16. PMID 21576639
- [Background] Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating MJ, Montserrat E, Rai KR, Kipps TJ; International Workshop on Chronic Lymphocytic Leukemia. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 guidelines. Blood. 2008 Jun 15;111(12):5446-56. doi: 10.1182/blood-2007-06-093906. Epub 2008 Jan 23. PMID 18216293
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Tsukasaki K, Hermine O, Bazarbachi A, Ratner L, Ramos JC, Harrington W Jr, O'Mahony D, Janik JE, Bittencourt AL, Taylor GP, Yamaguchi K, Utsunomiya A, Tobinai K, Watanabe T. Definition, prognostic factors, treatment, and response criteria of adult T-cell leukemia-lymphoma: a proposal from an international consensus meeting. J Clin Oncol. 2009 Jan 20;27(3):453-9. doi: 10.1200/JCO.2008.18.2428. Epub 2008 Dec 8. PMID 19064971